CLINICAL TRIAL: NCT04811417
Title: Frailty Assessment Among Kidney Transplant Candidates on the Waiting List
Brief Title: Frailty Assessment Among Kidney Transplant Candidates
Acronym: Mar-Kid
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, M José Pérez Sáez, Principal Investigator, Parc de Salut Mar
Other Study IDs: 2018/7798/I
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Frailty; Kidney Transplant; Complications
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is common among chronic kidney disease patients who are on the kidney transplant (KT) waiting list.

The aim of this study is to assess frailty according to different frailty tools among KT candidates and to establish potential biomarkers of frailty.

DETAILED DESCRIPTION:
This is an observational study where KT candidates will be assessed for frailty according to:

* Frailty Fried Phenotype and
* FRAIL scale

Sociodemographics and clinical variables will be collected and serum samples will be obtained in order to implement further studies regarding biomarkers of frailty..

ELIGIBILITY:
Inclusion Criteria:

* KT candidates accepted for the KT waiting list

Exclusion Criteria:

* No willing for participating
* Difficulty in understanding Spanish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: KT candidates (>18 years-old) accepted for the KT waiting list and willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of frailty among KT candidates | 2015-2020
  Prevalence of frailty according FRIED and FRAIL scale
Biomarkers of frailty among KT candidates | 2015-2020
  Serum samples for biomarkers

IPD SHARING:
Plan to Share IPD: No